CLINICAL TRIAL: NCT06551246
Title: Efficacy of Solifenacin, Mirabegron and Combination Therapy in Children With Overactive Bladder and Daytime Urinary Incontinence (BeDry)
Brief Title: Efficacy of Solifenacin, Mirabegron and Combination Therapy in Children With Daytime Urinary Incontinence (BeDry)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeDry
Record Dates: First submitted 2024-06-25; First posted 2024-08-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence in Children
Keywords: Urinary incontinence; Daytime urinary incontinence; Overactive bladder; Children; Solifenacin; Mirabegron
MeSH Terms: conditions — Urinary Incontinence; Diurnal Enuresis; Urinary Bladder, Overactive | interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Intervention Model Description: Children aged 5-14 years diagnosed with daytime urinary incontinence refractory to standard urotherapy will be randomized to four treatment groups, randomization 1:1:1:1.
Who Masked: Investigator
Masking Description: The study is single-blinded, and the study subject will receive medication delivered from the study site. The investigator does not know which treatment the individual participant receives. Participants will be informed that they are not allowed to reveal the blinded investigator the study medication, and an unblinded nurse will guide and answer questions to participants in case of dose titration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Solifenacin 5 mg + add-on solifenacin 5 mg (Experimental): Group 1A: Solifenacin 5 mg for 6 weeks, and if non-complete response after 6 weeks add-on solifenacin 5 mg for 12 weeks.
  Interventions: Drug: Solifenacin
- Solifenacin 5 mg + add-on mirabegron 25 mg (Experimental): Group 1B: Solifenacin 5 mg for 6 weeks, and if non-complete response after 6 weeks add-on mirabegron 25 mg for 12 weeks.
  Interventions: Drug: Solifenacin; Drug: Mirabegron
- Mirabegron 25 mg + ad-on mirabegron 25 mg (Experimental): Group 2A: Mirabegron 25 mg for 6 weeks, and if non-complete response after 6 weeks add-on mirabegron 25 mg for 12 weeks.
  Interventions: Drug: Mirabegron
- Mirabegron 25 mg + add-on solifenacin 5 mg (Experimental): Group 2B: Mirabegron 25 mg for 6 weeks, and if non-complete response after 6 weeks add-on solifenacin 5 mg for 12 weeks.
  Interventions: Drug: Solifenacin; Drug: Mirabegron

INTERVENTIONS:
Drug: Solifenacin — According to randomization.
  Arms: Mirabegron 25 mg + add-on solifenacin 5 mg; Solifenacin 5 mg + add-on mirabegron 25 mg; Solifenacin 5 mg + add-on solifenacin 5 mg
Drug: Mirabegron — According to randomization.
  Arms: Mirabegron 25 mg + ad-on mirabegron 25 mg; Mirabegron 25 mg + add-on solifenacin 5 mg; Solifenacin 5 mg + add-on mirabegron 25 mg

SUMMARY:
The primary objective is to evaluate if (1) combination therapy of solifenacin and mirabegron in low doses is superior to monotherapy of solifenacin in high dose and if (2) combination therapy of mirabegron and solifenacin in low doses is superior to monotherapy of mirabegron in high dose in treatment of daytime urinary incontinence among children aged 5 to 14 years who are none complete responders to respectively monotherapy of solifenacin in low dose or monotherapy of mirabegron in low dose.

In total, 236 children diagnosed with daytime urinary incontinence will be randomized 1:1:1:1 to one of four treatment groups. Total pharmacological treatment period will be 18 weeks.

DETAILED DESCRIPTION:
Background: According to International Children's Continence Society, first-line treatment of children with daytime urinary incontinence is standard urotherapy, eventually followed by pharmacotherapy of anticholinergics. The effect of medical treatment is sparsely investigated and primarily in non-randomized trials.

Objectives: The primary objective is to evaluate if (1) combination therapy of solifenacin and mirabegron in low doses is superior to monotherapy of solifenacin in high dose and if (2) combination therapy of mirabegron and solifenacin in low doses is superior to monotherapy of mirabegron in high dose in treatment of daytime urinary incontinence among children aged 5 to 14 years who are none complete responders to respectively monotherapy of solifenacin in low dose or monotherapy of mirabegron in low dose.

The secondary objective is to evaluate the treatment response of combination therapy of solifenacin and mirabegron in low doses, monotherapy in high dose and monotherapy in low doses as supplementary comparisons. Additionally, the secondary objective is to evaluate side effects, safety, and tolerability of the medical treatment as well as the effect of treatment on well-being and quality of life.

Study design: The BeDry study is designed as a multicenter, randomized, single-blinded, controlled clinical trial. Included children will be randomized 1:1:1:1 to one of four treatment groups. Children aged 5-14 years diagnosed with daytime urinary incontinence refractory to standard urotherapy will be randomized. Initially two groups will receive solifenacin 5 mg and two groups will receive mirabegron 25 mg. After 6 weeks, non-complete respondsers will receive add-on treatment according to their primary randomization group; group 1A will reviece solifenacin 5 mg and add-on solifenacin 5 mg, group 1B will receive solifenacin 5 mg and add-on mirabegron 25 mg, group 2A will receive mirabegron 25 mg and add-on mirabegron 25 mg, group 2B will receive mirabegron 25 mg and add-on solifenacin 5 mg. Total treatment period will be 18 weeks. The primary endpoint measure is treatment response assessed by change from visit 2 to end of study, according to number of wet days pr. 7 days by DryPie.

Perspectives: The trial has the potential to optimize medical treatment of children with daytime urinary incontinence, to shorten the treatment period, diminish side effects and minimized unnecessary medical expenses.

Ethics: All pharmacological side effects will be handled in accordance with the Danish legislation. No risk or unknown side effects are expected to urotherapy, medical treatment or withdrawal. No risks are expected by the clinical examination and paraclinical measurements. The therapeutic potential for future patients justifies the project to be carried out. Participation in this study will not lead to any disadvantages for the patient in their treatment. The study will be conducted in accordance with the protocol, applicable regulatory requirements according to Good Clinical Practice and the ethical principles of the Declaration of Helsinki. The study is approved by the authorities. Significant additions or changes to the protocol may be conducted after the application for amendment is approved by the Regulatory Authority and the Ethics Committee. Information regarding the participants is protected according to the General Data Protection Regulation and the actual law. The study is registered at the research inventory of the Regions of Denmark (1-16-02-210-24) and at Aarhus University (ARG-2024-731-23829). The study is registered and authorized at CTIS (EU CT 2023-510187-13-00).

ELIGIBILITY:
Inclusion Criteria:

1. The participants custody holder(s) must voluntarily sign and date an informed consent prior to initiation of any study specific procedures.
2. Age 5 to 14 years (inclusive) at the time of inclusion.
3. Overactive bladder as per International Children's Continence Society criteria
4. At least 2 daytime urinary incontinence episodes per week
5. Inadequate effect of at least 4 weeks urotherapy (non-pharmacological treatment)
6. No previous treatment with solifenacin, mirabegron or bladder/sphincter botulinum toxin injections
7. No current constipation as per ROME IV criteria or fecal incontinence (laxative treatment is accepted)
8. Per investigator's judgment, the participant can swallow or can learn to swallow study medication

Exclusion Criteria:

1. Inability of the patent(s) or legal guardian(s) to understand the Danish written and oral information
2. Known or suspected hypersensitivity to study medication
3. Any contraindication to the use of the study medication
4. Known urogenital anatomical abnormalities affecting lower urinary tract function
5. Known kidney or bladder stones
6. Known diabetes insipidus
7. Ongoing symptomatic urinary tract infection
8. Recurrent urinary tract infection or ongoing prophylactic antibiotic treatment
9. Known QTc prolongation, QTc >460 ms, or risk of QTc prolongation (hypokalaemia, exercise-induced syncope, or familial long QT syndrome)
10. Other significant electrocardiogram abnormalities
11. Known hypertension
12. ≤3 daily voiding, evaluated by 48-hour frequency-volume chart
13. Uroflowmetry suggestive of other pathology than overactive bladder (staccato-shaped, interrupted-shaped, or plateau-shaped curve)
14. Post-void residual >50 ml after double voiding
15. Dipstick haematuria (≥2+ erythrocytes) or macroscopic haematuria
16. Pregnancy or breastfeeding
17. Female subjects of childbearing potential
18. Ongoing constipation according to Rome IV-criteria which is intractable to medication or fecal incontinence
19. Inability to swallow study medication
20. Use of any medication during study period, except permitted medication

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment response | From study week 6 and through study completion, an average of 18 weeks in total
  Assesed by change in number of wetdays pr. 7 days by DryPie

SECONDARY OUTCOMES:
Treatment response | From date of randomization until study completion, an average of 18 weeks in total
  Assesed by change in number of wetdays pr. 7 days by DryPie
Inconcintnence severity score | From date of randomization until study completion, an average of 18 weeks in total
  Assesed by DryPie (scoring from 0 to 21, in which the higher score means severe incontinence)
Urge severity | From date of randomization until study completion, an average of 18 weeks in total
  Quantified by Bower VAS Urgency Scheme (scoring from 0 to 10, in which the higher score means servere urge)
Maximum voided volume (ml) | From date of randomization until study completion, an average of 18 weeks in total
  48-hour frequency-volume chart
Age standardized maximum voided volume (ml) | From date of randomization until study completion, an average of 18 weeks in total
  Maximum voided volume as a percent of expected bladder capacity
Average voided volume (ml) | From date of randomization until study completion, an average of 18 weeks in total
  48-hour frequency-volume chart
Miction frequency | From date of randomization until study completion, an average of 18 weeks in total
  48-hour frequency-volume chart
Pediatric incontinence questionnaire total score | From date of randomization until study completion, an average of 18 weeks in total
  20-item questionnaire (scoring from 0 to 4 on a Likert scale, with a total of 80 points in which the higher score, the greater impact of urinary incontinence of quality of life)
WHO-5 total score | From date of randomization until study completion, an average of 18 weeks in total
  5-item questionnaire (scoring from 0 to 5 on a Likert scale, with a total of 30 points in which the higher score, the greater impact of urinary incontinence of quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Luise Borch, MD, PhD, Study Director — Department of Pediatric and Adolescent Medicine, Gødstrup Hospital
Locations (5):
- Denmark (5):
  - Department of Pediatric and Adolescent Medicine, Aalborg University Hospital, Aalborg, Aalborg
  - Department of Pediatric and Adolescent Medicine, Aarhus University Hospital, Aarhus, Aarhus N
  - Department of Pediatric and Adolescent medicine, Esbjerg Hospital, Esbjerg, Esbjerg
  - Department of Pediatric and Adolescent Medicine, Gødstrup Hospital, Herning, Herning
  - Department of Pediatric and Adolescent Medicine, Kolding Hospital, Kolding, Kolding

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svendsen AM, Hagstrom S, Thorsteinsson K, Van Batavia J, Kamperis K, Olesen AE, Borch L. Efficacy of Solifenacin, Mirabegron, and Combination Therapy in Children With Daytime Urinary Incontinence (BeDry): Protocol for a Randomized Single-Blinded Controlled Trial. JMIR Res Protoc. 2025 Jun 26;14:e63588. doi: 10.2196/63588. PMID 40570329